CLINICAL TRIAL: NCT02184143
Title: Comparative Effectiveness of Postoperative Management for Degenerative Spinal Conditions
Brief Title: Postoperative Management for Degenerative Spinal Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Kristin Archer, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 140057
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-06

CONDITIONS: Spinal Degenerative Disorder
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBPT intervention (Experimental): CBPT program consisting of weekly phone calls.
  Interventions: Behavioral: CBPT
- Education intervention (Active Comparator): Education program consisting of weekly phone calls.
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: CBPT — Changing Behavior through Physical Therapy (CBPT) is a cognitive-behavioral based self-management program.
  Arms: CBPT intervention
Other: Education — Patient education
  Arms: Education intervention

SUMMARY:
The overall objective of this study is to conduct a two-group randomized control trial (RCT) to compare which of two treatments provided by telephone - a cognitive-behavioral based physical therapy (CBPT) program focusing on self-management strategies or an education program about postoperative recovery - are more effective for improving patient-centered outcomes in older adults recovering from lumbar spine surgery for degenerative conditions. Our central hypothesis is that the CBPT intervention focusing on self-management will decrease pain and disability and improve general health, physical activity and physical function in community-dwelling adults undergoing spine surgery, through reductions in fear of movement and increases in pain self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Radiographic evidence of lumbar spinal stenosis secondary to degenerative changes
2. Surgical treatment of a lumbar degenerative condition (spinal stenosis, spondylosis with or without myelopathy, and degenerative spondylolisthesis) using laminectomy with or without arthrodesis procedures
3. English speaking due to feasibility of employing study personnel to deliver and assess the study intervention
4. Age older than 21 years (younger individuals do not typically have a lumbar degenerative condition).

Exclusion Criteria:

1. Patients having microsurgical techniques as the primary procedure, such as an isolated laminotomy or microdiscectomy (individuals having these minimally invasive surgical techniques tend to have a less severe case of lumbar degeneration and a shorter recovery time than individuals having arthrodesis or laminectomy without arthrodesis)
2. Patients having surgery for spinal deformity as the primary indication (patients with spinal deformity as the primary spinal disorder tend to have a different recovery trajectory compared to the inclusion population)
3. Patients having surgery secondary to pseudarthrosis, trauma, infection, or tumor
4. Presence of back and/or lower extremity pain < 3 months indicating no history of chronic pain
5. History of neurological disorder or disease, resulting in moderate to severe movement dysfunction. Including but not limited to Parkinson's disease, Multiple Sclerosis, Epilepsy, Brain tumors, Huntington's disease, Alzheimer's disease, Muscular Dystrophy, Stroke, Autonomic Nervous System disorders, Traumatic Brain Injury, Cerebral Palsy, and Amyotrophic Lateral Sclerosis
6. Presence of schizophrenia or other psychotic disorder, including but not limited to Brief Psychotic disorder and Delusional disorder
7. Patients not able to return to clinic for standard follow-up visits with surgeon due to time and travel limitation
8. Patients having surgery under a workman's compensation claim
9. Unable to provide a stable address and access to a telephone indicating the inability to participate in either the telephone-based CBPT or education program.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2014-08; Primary Completion 2017-11 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin R Archer, PT, PhD, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Background] Archer KR, Motzny N, Abraham CM, Yaffe D, Seebach CL, Devin CJ, Spengler DM, McGirt MJ, Aaronson OS, Cheng JS, Wegener ST. Cognitive-behavioral-based physical therapy to improve surgical spine outcomes: a case series. Phys Ther. 2013 Aug;93(8):1130-9. doi: 10.2522/ptj.20120426. Epub 2013 Apr 18. PMID 23599351
- [Background] Archer KR, Devin CJ, Vanston SW, Koyama T, Phillips SE, Mathis SL, George SZ, McGirt MJ, Spengler DM, Aaronson OS, Cheng JS, Wegener ST. Cognitive-Behavioral-Based Physical Therapy for Patients With Chronic Pain Undergoing Lumbar Spine Surgery: A Randomized Controlled Trial. J Pain. 2016 Jan;17(1):76-89. doi: 10.1016/j.jpain.2015.09.013. Epub 2015 Oct 23. PMID 26476267
- [Derived] Archer KR, Coronado RA, Haug CM, Vanston SW, Devin CJ, Fonnesbeck CJ, Aaronson OS, Cheng JS, Skolasky RL, Riley LH 3rd, Wegener ST. A comparative effectiveness trial of postoperative management for lumbar spine surgery: changing behavior through physical therapy (CBPT) study protocol. BMC Musculoskelet Disord. 2014 Oct 1;15:325. doi: 10.1186/1471-2474-15-325. PMID 25273991

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 838 participants assessed for eligibility. Of these 838, 513 participants were excluded. Of these 513 who were excluded, 222 did not meet inclusion criteria, 268 declined to participate, 23 were assessed too close to surgery to complete a preoperative assessment.
Pre-assignment Details: 248 participants were consented, enrolled, and randomized.
Groups:
- CBPT Intervention: Subjects participate in the cognitive behavioral physical therapy (CBPT) program focusing on a patient-oriented self-management approach to reduce pain and disability and improve physical activity and function, through reductions in fear of movement and increases in self-efficacy. Program consists of six weekly telephone sessions with a trained physical therapist. The first session is 45 minutes and the remaining 5 sessions are 30 minutes. Each subject received a binder to follow along with study therapist.
- Education Intervention: Subjects participate in an education program focusing on postoperative recovery. Sessions address benefits of physical therapy, proper biomechanics after surgery, importance of daily exercise, ways to promote healing, stress reduction, sleep hygiene, energy management, communication with health providers, and preventing future injury. Treatment Group 2 is matched to the Treatment Group 1 in terms of session frequency, length and contact with the study therapist. Each subject received a binder to follow along with study therapist.
Period: Overall Study
Arm/Group | CBPT Intervention | Education Intervention
Started | 124 (124 participants randomized; 118 participant received intervention) | 124 (124 participants randomized; 121 received intervention)
Completed | 114 (114 patients completed PROs. 98 actigraph valid wear time.) | 117 (117 patients completed PROs. 100 actigraph valid wear time.)
Not Completed | 10 | 7
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Lost to Follow-up | 5 | 3
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- CBPT Intervention: Subjects participate in the cognitive behavioral physical therapy (CBPT) program focusing on a patient-oriented self-management approach to reduce pain and disability and improve physical activity and function, through reductions in fear of movement and increases in self-efficacy. Program consists of six weekly telephone sessions with a trained physical therapist. The first session is 45 minutes and the remaining 5 sessions are 30 minutes. Each subject will receive a binder to follow along with study therapist.
- Education Intervention: Subjects participate in an education program focusing on postoperative recovery. Sessions address benefits of physical therapy, proper biomechanics after surgery, importance of daily exercise, ways to promote healing, stress reduction, sleep hygiene, energy management, communication with health providers, and preventing future injury. Treatment Group 2 is matched to the Treatment Group 1 in terms of session frequency, length and contact with the study therapist. Each subject will receive a binder to follow along with study therapist.
- Total: Total of all reporting groups
Arm/Group | CBPT Intervention | Education Intervention | Total
Number analyzed (Participants) | 124 | 124 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.94 (11.50) | 61.44 (12.22) | 62.19 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 66 | 126
  Male | 64 | 58 | 122
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 107 | 108 | 215
  Non-White | 17 | 16 | 33
Marital Status [Count of Participants; unit: Participants]
  Single | 16 | 7 | 23
  Married | 81 | 83 | 164
  Widowed | 9 | 13 | 22
  Divorced | 15 | 15 | 30
  Separated | 0 | 3 | 3
  Living with Partner | 3 | 3 | 6
Educational Level [Count of Participants; unit: Participants]
  Less than 12th grade | 5 | 3 | 8
  12th grade, diploma or GED | 26 | 32 | 58
  Some college, no degree | 33 | 43 | 76
  Associate degree | 16 | 11 | 27
  College degree | 24 | 19 | 43
  Graduate degree | 20 | 16 | 36
Insurance Status [Count of Participants; unit: Participants]
  Private | 57 | 68 | 125
  Public (i.e., Medicare, Medicaid) | 57 | 49 | 106
  Military health plan (i.e., TRICARE) | 10 | 7 | 17
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.18 (6.12) | 32.59 (7.01) | 32.39 (6.57)
Current tobacco use [Count of Participants; unit: Participants] | 18 | 21 | 39
Working status [Count of Participants; unit: Participants]
  Employed | 45 | 46 | 91
  Retired (not due to illness) | 41 | 41 | 82
  Disabled and/or retired due to illness | 35 | 31 | 66
  Looking for work | 1 | 0 | 1
  Elected not to work (e.g., Homemaker) | 0 | 5 | 5
  Attending School | 2 | 1 | 3
Pain duration [Median (Inter-Quartile Range); unit: months] | 16.5 [8.00 to 57.00] | 24 [11.25 to 48.00] | 23 [9.25 to 48.00]
Prior spinal surgery [Count of Participants; unit: Participants] | 32 | 42 | 74
Comorbidities [Count of Participants; unit: Participants]
  None | 53 | 64 | 117
  One | 49 | 38 | 87
  Two or more | 22 | 22 | 44
Narcotics: yes [Count of Participants; unit: Participants] | 49 | 43 | 92
Surgery type [Count of Participants; unit: Participants]
  Laminectomy without fusion | 51 | 33 | 84
  Laminectomy with fusion | 73 | 91 | 164
Spinal Levels [Count of Participants; unit: Participants]
  One | 56 | 55 | 111
  Two | 47 | 45 | 92
  Three or more | 21 | 24 | 45
Revision Surgery [Count of Participants; unit: Participants] | 17 | 18 | 35
Length of Stay (LOS) [Mean (Standard Deviation); unit: days] | 3.01 (1.82) | 3.6 (3.32) | 3.31 (2.69)
Discharge location [Count of Participants; unit: Participants]
  Home | 87 | 88 | 175
  Home with services | 20 | 14 | 34
  Skilled nursing facility | 3 | 10 | 13
  Inpatient rehabilitation facility | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Oswestry Disability Index (ODI)
Description: The ODI measures disease-specific disability on a scale from 0 to 100, with higher scores indicating worse disability.
Time Frame: Up to 12 months.
Population: Number analyzed indicate the number of participants who completed the measure at each time point.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CBPT Intervention | Education Intervention
Number analyzed (Participants) | 124 | 124
units on a scale
  Preoperative: number analyzed (Participants) | 118 | 120
  Preoperative | 43.6 [40.88 to 46.33] | 45.46 [42.80 to 48.11]
  Baseline (6 weeks): number analyzed (Participants) | 123 | 124
  Baseline (6 weeks) | 31.31 [27.98 to 34.65] | 31.19 [28.16 to 34.23]
  6 Months: number analyzed (Participants) | 117 | 119
  6 Months | 24.06 [20.68 to 27.43] | 24.33 [21.34 to 27.32]
  12 Months: number analyzed (Participants) | 114 | 117
  12 Months | 23.37 [19.92 to 26.81] | 26.17 [22.99 to 29.35]

2. Primary Outcome: Brief Pain Inventory (BPI)
Description: The BPI measures pain from 0 to 10, with higher scores indicating a worse outcome
Time Frame: Up to 12 months after spine surgery
Population: Number analyzed indicate the number of participants who completed the measure at each time point.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CBPT Intervention | Education Intervention
Number analyzed (Participants) | 124 | 124
units on a scale
  Back Pain: Preoperative: number analyzed (Participants) | 120 | 123
  Back Pain: Preoperative | 6.79 [6.4 to 7.18] | 6.64 [6.22 to 7.06]
  Back Pain: 6 Week: number analyzed (Participants) | 123 | 124
  Back Pain: 6 Week | 3.15 [2.69 to 3.6] | 3.14 [2.74 to 3.54]
  Back Pain: 6 Month: number analyzed (Participants) | 116 | 119
  Back Pain: 6 Month | 2.82 [2.39 to 3.24] | 2.69 [2.28 to 3.1]
  Back Pain: 12 Month: number analyzed (Participants) | 114 | 115
  Back Pain: 12 Month | 2.95 [2.46 to 3.43] | 2.83 [2.38 to 3.27]
  Leg Pain: Preoperative: number analyzed (Participants) | 119 | 122
  Leg Pain: Preoperative | 6.63 [6.2 to 7.06] | 6.38 [5.92 to 6.83]
  Leg Pain: 6 Week: number analyzed (Participants) | 123 | 124
  Leg Pain: 6 Week | 2.32 [1.88 to 2.75] | 2.35 [1.9 to 2.81]
  Leg Pain: 6 Month: number analyzed (Participants) | 116 | 119
  Leg Pain: 6 Month | 2.23 [1.77 to 2.69] | 2.45 [1.98 to 2.91]
  Leg Pain: 12 Month: number analyzed (Participants) | 114 | 115
  Leg Pain: 12 Month | 2.35 [1.87 to 2.83] | 2.81 [2.28 to 3.34]

3. Primary Outcome: 12-Item Short Form Health Survey (SF-12)
Description: The SF-12 is a measure of general physical and mental health. The SF-12 is scored from 0 to 100, with higher scores indicating better health.
Time Frame: Up to 12 months after spine surgery
Population: Number analyzed indicate the number of participants who completed the measure at each time point.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CBPT Intervention | Education Intervention
Number analyzed (Participants) | 124 | 124
units on a scale
  Physical Health: Preoperative: number analyzed (Participants) | 117 | 119
  Physical Health: Preoperative | 27.84 [26.19 to 29.5] | 27.8 [26.22 to 29.38]
  Physical Health: 6 Week: number analyzed (Participants) | 123 | 124
  Physical Health: 6 Week | 33.49 [31.61 to 35.36] | 33.55 [31.99 to 35.1]
  Physical Health: 6 Month: number analyzed (Participants) | 116 | 119
  Physical Health: 6 Month | 39.31 [37.11 to 41.5] | 38.81 [36.86 to 40.77]
  Physical Health: 12 Month: number analyzed (Participants) | 114 | 115
  Physical Health: 12 Month | 39.25 [36.82 to 41.69] | 37.43 [35.21 to 39.64]
  Mental Health: Preoperative: number analyzed (Participants) | 117 | 118
  Mental Health: Preoperative | 49.69 [47.55 to 51.84] | 48.54 [46.23 to 50.86]
  Mental Health: 6 Week: number analyzed (Participants) | 123 | 124
  Mental Health: 6 Week | 52.27 [50.25 to 54.29] | 51.89 [49.75 to 54.02]
  Mental Health: 6 Month: number analyzed (Participants) | 116 | 119
  Mental Health: 6 Month | 54.02 [52.46 to 55.58] | 52.94 [50.84 to 55.03]
  Mental Health: 12 Month: number analyzed (Participants) | 114 | 115
  Mental Health: 12 Month | 53.86 [52.01 to 55.71] | 53.23 [51.38 to 55.08]

4. Secondary Outcome: Physical Activity
Description: Physical activity measured by a commercially available movement accelerometer
Time Frame: Up to 12 months after spine surgery
Population: Number analyzed indicate the number of participants who completed the measure at each time point.
Measure: Mean (95% Confidence Interval); unit: Mean Activity Counts/Minute
Arm/Group | CBPT Intervention | Education Intervention
Number analyzed (Participants) | 124 | 124
Mean Activity Counts/Minute
  Mean Activity Counts/Minute: 6 weeks: number analyzed (Participants) | 106 | 109
  Mean Activity Counts/Minute: 6 weeks | 432.17 [390.69 to 473.66] | 421.77 [386.08 to 457.45]
  Mean Activity Counts/Minute: 6 months: number analyzed (Participants) | 101 | 105
  Mean Activity Counts/Minute: 6 months | 484.29 [443.08 to 525.51] | 487.93 [440.90 to 534.97]
  Mean Activity Counts/Minute: 12 months: number analyzed (Participants) | 98 | 100
  Mean Activity Counts/Minute: 12 months | 474.29 [427.66 to 520.92] | 480.42 [440.48 to 520.36]

ADVERSE EVENTS:
Time Frame: Adverse event data collected over 12 months.
Arm/Group | CBPT Intervention | Education Intervention
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/124
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/124
Other Adverse Events (participants affected / at risk) | 0/124 | 0/124

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT02184143/Prot_SAP_000.pdf